CLINICAL TRIAL: NCT04695379
Title: Follow-up of a Cohort of Patients With Myasthenic Syndrome and COVID-19 Infection: Consequences on the Severity of Myasthenic Syndrome and Reciprocal Impact of the Two Pathologies on Their Respective Treatments
Brief Title: Follow-up of a Cohort of Patients With Myasthenic Syndrome and COVID-19 Infection
Acronym: CO-MY-COVID
Status: Completed | Type: Observational
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Other Study IDs: CHUBX 2020/17
Record Dates: First submitted 2020-12-31; First posted 2021-01-05 (Actual); Last update posted 2023-10-06 (Actual); Status verified 2023-10

CONDITIONS: Myasthenia Gravis
Keywords: COVID-19; Neuromuscular Diseases
MeSH Terms: conditions — Myasthenia Gravis; COVID-19; Neuromuscular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Coronavirus disease 2019 (COVID-19), declared by the World Health Organization (WHO) as a "public health emergency of international concern" (January 31, 2020), has posed a significant threat to global health. This infectious disease, caused by the 'severe acute respiratory syndrome coronavirus-2'(SARS-CoV-2), was first reported in China at the end of 2019. As other coronaviruses, SARS-CoV-2 primarily targets the human respiratory system. The most common symptoms are fever, fatigue, and dry cough. During the second week of the disease, part of patients may progress to shortness of breath, then hypoxemia and severe pneumonia. Acute respiratory distress syndrome (ARDS), linked to some risk factors such as advanced age and underlying comorbidities (hypertension, diabetes, cardiovascular disease, and cerebrovascular disease), may be fatal and needs early supportive therapy and monitoring.

Some patients with COVID-19 experienced neurological complications including headache, dizziness, hypogeusia and/or anosmia, altered level of consciousness, strokes, seizures, and ataxia, less frequently neuromuscular disorders (NMD) such as acute inflammatory polyradiculoneuropathy. Among NMD, myasthenia gravis (MG) patients, particularly susceptible to infections causing crises, could be of special risk of COVID-19 ARDS. Some general recommendations were established for the management of NMD during the COVID-19 pandemic,with also specific recommendations for MG. However, only data on a small number of patients who were managed in hospital are currently available;in addition, only two cases of myasthenic crisis following COVID-19 were reported. For this reason, the French neuromuscular rare disease network (FILNEMUS: 'FILière NEuroMUSculaire') has created the 'CO-MY-COVID register' to describe the clinical course and prognosis of patients with COVID-19 and pre-existing myasthenic syndrome.

DETAILED DESCRIPTION:
Coronavirus disease 2019 (COVID-19), declared by the World Health Organization (WHO) as a "public health emergency of international concern" (January 31, 2020), has posed a significant threat to global health. This infectious disease, caused by the 'severe acute respiratory syndrome coronavirus-2'(SARS-CoV-2), was first reported in China at the end of 2019. Nowadays, with the exception of Antarctica, COVID-19 is a worldwide pandemic that continues to spread around the world (8,065,966 known cases and 437,604 deaths in June 16, 2020; https://gisanddata.maps.arcgis.com/). As other coronaviruses, SARS-CoV-2 primarily targets the human respiratory system. Its most convincing mode of transmission is inhalation of infectious aerosols or direct contact of infected people's droplets. The most common symptoms are fever, fatigue, and dry cough. During the second week of the disease, part of patients may progress to shortness of breath, then hypoxemia and severe pneumonia. Acute respiratory distress syndrome (ARDS), linked to some risk factors such as advanced age and underlying comorbidities (hypertension, diabetes, cardiovascular disease, and cerebrovascular disease), may be fatal and needs early supportive therapy and monitoring.

Some patients with COVID-19 experienced neurological complications including headache, dizziness, hypogeusia and/or anosmia, altered level of consciousness, strokes, seizures, and ataxia, less frequently neuromuscular disorders (NMD) such as acute inflammatory polyradiculoneuropathy. Among NMD, myasthenia gravis (MG) patients, particularly susceptible to infections causing crises, could be of special risk of COVID-19 ARDS. Some general recommendations were established for the management of NMD during the COVID-19 pandemic,with also specific recommendations for MG. However, only data on a small number of patients who were managed in hospital are currently available;in addition, only two cases of myasthenic crisis following COVID-19 were reported. For this reason, the French neuromuscular rare disease network (FILNEMUS: 'FILière NEuroMUSculaire') has created the 'CO-MY-COVID register' to describe the clinical course and prognosis of patients with COVID-19 and pre-existing myasthenic syndrome.

ELIGIBILITY:
Inclusion Criteria:

* 1. Child or adult patients, living or deceased, presenting or having presented a myasthenic syndrome and a COVID-19 infection 2. Myasthenic syndrome is established by:

  * Either the presence of a specific antibody
  * Either the presence of specific electrophysiological abnormalities
  * Either an evocative symptomatology improved by a therapeutic test with an acetylcholinesterase inhibitor
  * Either one or two pathogenic mutation (s) in a gene involved in congenital myasthenic syndromes (dominant or recessive disease).

    3. COVID-19 infection is established by
  * Either a positive PCR test
  * Or a specific chest scanner
  * Either a positive serology
  * Either a clinical syndrome of COVID-19, validated by a committee of experts. 4. Patients affiliated or beneficiaries of a social security scheme 5. For living patients: patients who have been informed of the study and have not exercised their right of opposition or parents or holders of parental authority who have been informed of the study and have not exercised their right opposition.

For deceased patients: beneficiaries or parents / holders of parental authority having been informed of the study and not having exercised their right of objection.

Exclusion Criteria:

1. Persons placed under judicial protection

Ages: 1 Year to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Child or adult patients, living or deceased, presenting or having presented a myasthenic syndrome and a COVID-19 infection
Sampling Method: Non-Probability Sample
Enrollment: 34 (Actual)
Dates: Start 2020-04-27 (Actual); Primary Completion 2020-06-18 (Actual); Study Completion 2020-06-18 (Actual)

PRIMARY OUTCOMES:
Severity of Myasthenia Gravis evaluated by the Myasthenia Gravis of America (MGFA) score | 1 month after the inclusion visit
  The severity of MG is measured by using the MGFA (Myasthenia Gravis Foundation of America) classification, giving the status of 'MG-improvement' (when the scores decreased or remained stable) or 'MG-worsening' (when the scores increased) (Jaretzki A, 3rd, Barohn RJ, Ernstoff RM, et al. Myasthenia gravis: recommendations for clinical research standards. Task Force of the Medical Scientific Advisory Board of the Myasthenia Gravis Foundation of America. Neurology 2000;55:16-23.)

SECONDARY OUTCOMES:
Severity of Myasthenia Gravis evaluated by the Myasthenia Gravis of America (MGFA) score | at inclusion (at the time of the COVID-19 diagnosis)
  The severity of MG is measured by using the MGFA (Myasthenia Gravis Foundation of America) classification, giving the status of 'MG-improvement' (when the scores decreased or remained stable) or 'MG-worsening' (when the scores increased) (Jaretzki A, 3rd, Barohn RJ, Ernstoff RM, et al. Myasthenia gravis: recommendations for clinical research standards. Task Force of the Medical Scientific Advisory Board of the Myasthenia Gravis Foundation of America. Neurology 2000;55:16-23.)
Severity of Myasthenia Gravis evaluated by the variation of the Myasthenia Gravis of America (MGFA) score | 3 months after the inclusion visit
  The severity of MG is measured by using the MGFA (Myasthenia Gravis Foundation of America) classification, giving the status of 'MG-improvement' (when the scores decreased or remained stable) or 'MG-worsening' (when the scores increased) (Jaretzki A, 3rd, Barohn RJ, Ernstoff RM, et al. Myasthenia gravis: recommendations for clinical research standards. Task Force of the Medical Scientific Advisory Board of the Myasthenia Gravis Foundation of America. Neurology 2000;55:16-23.)
Severity of Myasthenia Gravis evaluated by the variation of the Myasthenia Gravis of America (MGFA) score | 6 months after the inclusion visit
  The severity of MG is measured by using the MGFA (Myasthenia Gravis Foundation of America) classification, giving the status of 'MG-improvement' (when the scores decreased or remained stable) or 'MG-worsening' (when the scores increased) (Jaretzki A, 3rd, Barohn RJ, Ernstoff RM, et al. Myasthenia gravis: recommendations for clinical research standards. Task Force of the Medical Scientific Advisory Board of the Myasthenia Gravis Foundation of America. Neurology 2000;55:16-23.)
The autonomy of the patients evaluated with the MG-ADL (Myasthenia Gravis-Activities of Daily Living) scale | at inclusion (at the time of the COVID-19 diagnosis)
  The Myasthenia Gravis-specific Activities of Daily Living scale consists of the assessment of 8 parameters: speaking, chewing, swallowing, breathing, self-care activities (brushing the teeth or combing the hair), simple physical activities (getting up from a chair), double vision and eye lid dropping. Each parameter is subjected to assessment depending on the degree of symptoms intensification, awarding points from 0 to 3 points. The maximum number a patient may receive is 24 points. The higher the score of points, the bigger limitations of the patient in everyday life activities caused by intensification of myasthenia gravis (Wolfe GI, Herbelin L, Nations SP, Foster B, Bryan WW, Barohn RJ. Myasthenia gravis activities of daily living profile. Neurology 1999;52:1487-1489.)
The autonomy of the patients evaluated with the MG-ADL (Myasthenia Gravis-Activities of Daily Living) scale | 1 month after the inclusion visit
  The Myasthenia Gravis-specific Activities of Daily Living scale consists of the assessment of 8 parameters: speaking, chewing, swallowing, breathing, self-care activities (brushing the teeth or combing the hair), simple physical activities (getting up from a chair), double vision and eye lid dropping. Each parameter is subjected to assessment depending on the degree of symptoms intensification, awarding points from 0 to 3 points. The maximum number a patient may receive is 24 points. The higher the score of points, the bigger limitations of the patient in everyday life activities caused by intensification of myasthenia gravis (Wolfe GI, Herbelin L, Nations SP, Foster B, Bryan WW, Barohn RJ. Myasthenia gravis activities of daily living profile. Neurology 1999;52:1487-1489.)
The autonomy of the patients evaluated with the MG-ADL (Myasthenia Gravis-Activities of Daily Living) scale | 3 months after the inclusion visit
  The Myasthenia Gravis-specific Activities of Daily Living scale consists of the assessment of 8 parameters: speaking, chewing, swallowing, breathing, self-care activities (brushing the teeth or combing the hair), simple physical activities (getting up from a chair), double vision and eye lid dropping. Each parameter is subjected to assessment depending on the degree of symptoms intensification, awarding points from 0 to 3 points. The maximum number a patient may receive is 24 points. The higher the score of points, the bigger limitations of the patient in everyday life activities caused by intensification of myasthenia gravis (Wolfe GI, Herbelin L, Nations SP, Foster B, Bryan WW, Barohn RJ. Myasthenia gravis activities of daily living profile. Neurology 1999;52:1487-1489.)
The autonomy of the patients evaluated with the MG-ADL (Myasthenia Gravis-Activities of Daily Living) scale | 6 months after the inclusion visit
  The Myasthenia Gravis-specific Activities of Daily Living scale consists of the assessment of 8 parameters: speaking, chewing, swallowing, breathing, self-care activities (brushing the teeth or combing the hair), simple physical activities (getting up from a chair), double vision and eye lid dropping. Each parameter is subjected to assessment depending on the degree of symptoms intensification, awarding points from 0 to 3 points. The maximum number a patient may receive is 24 points. The higher the score of points, the bigger limitations of the patient in everyday life activities caused by intensification of myasthenia gravis (Wolfe GI, Herbelin L, Nations SP, Foster B, Bryan WW, Barohn RJ. Myasthenia gravis activities of daily living profile. Neurology 1999;52:1487-1489.)
Risk factors for severe forms of COVID-19 | at inclusion (at the time of the COVID-19 diagnosis)
  Risk factors for severe forms of COVID-19 are the following: age>65, 'obesity' (body mass index (, BMI), >30), 'chronic obstructive pulmonary disease' (COPD), 'obstructive sleep apnea syndrome' (OSAS), 'noninvasive ventilation' (NIV), 'arterial hypertension' , 'diabetes' and 'others'
Treatments for MG at the time of the diagnosis of COVID-19 | at inclusion (at the time of the COVID-19 diagnosis)
  Treatments for MG at the time of the diagnosis of COVID-19 are grouped into six categories: 'acetylcholinesterase inhibitors' (Ach-inh), 'corticosteroids', 'immunosuppressants', 'intravenous immunoglobulins' (IVIg) or 'subcutaneous immunoglobulins' (SCIg), 'plasmapheresis' (PLEX) and 'others
Diagnosis of COVID-19 | at inclusion (at the time of the COVID-19 diagnosis)
  The diagnosis of COVID-19 is considered as 'definite' if confirmed by a positive SARS-CoV-2 PCR (polymerase chain reaction) test and/or SARS-CoV-2 serology. The diagnosis of COVID-19 is considered 'probable' if: (i) the patient presented a viral syndrome and (ii) had contact with a confirmed patient considered to have a definite diagnosis of COVID-19 or had specific signs (anosmia, agueusia, skin signs) or had suggestive abnormalities on thoracic CT-scan.
Severity of COVID-19 | at inclusion (at the time of the COVID-19 diagnosis)
  The global severity of COVID-19 was based on the location of management of the patient during COIVD-19: 'home', 'medical unit' ('MU'), 'intensive care unit' ('ICU').
Treatments for MG during and after COVID-19 | 1 month after the inclusion visit
  Treatments for MG at the time of the diagnosis of COVID-19 are grouped into six categories: 'acetylcholinesterase inhibitors' (Ach-inh), 'corticosteroids', 'immunosuppressants', 'intravenous immunoglobulins' (IVIg) or 'subcutaneous immunoglobulins' (SCIg), 'plasmapheresis' (PLEX) and 'others
Treatments for MG during and after COVID-19 | 3 months after the inclusion visit
  Treatments for MG at the time of the diagnosis of COVID-19 are grouped into six categories: 'acetylcholinesterase inhibitors' (Ach-inh), 'corticosteroids', 'immunosuppressants', 'intravenous immunoglobulins' (IVIg) or 'subcutaneous immunoglobulins' (SCIg), 'plasmapheresis' (PLEX) and 'others
Treatments for MG during and after COVID-19 | 6 months after the inclusion visit
  Treatments for MG at the time of the diagnosis of COVID-19 are grouped into six categories: 'acetylcholinesterase inhibitors' (Ach-inh), 'corticosteroids', 'immunosuppressants', 'intravenous immunoglobulins' (IVIg) or 'subcutaneous immunoglobulins' (SCIg), 'plasmapheresis' (PLEX) and 'others

CONTACTS AND LOCATIONS:
Overall Officials: Guilhem SOLE, MD, Principal Investigator — Université Hospital, Bordeaux
Locations (10):
- France (10):
  - CHU d'Angers, Angers
  - CHU de Bordeaux, Bordeaux
  - Hospices Civils de Lyon, Bron
  - APHP - Hopital Raymond Poincarré, Garches
  - CHRU de Lille, Lille
  - Assistance Publique Hôpitaux de Marseille, Marseille
  - CHU de Nantes, Nantes
  - APHP GH Pitié Salpétrière, Paris
  - CHU de Strasbourg, Strasbourg
  - CHU de Toulouse, Toulouse